CLINICAL TRIAL: NCT01672411
Title: Predictive Value of Prostate-specific Antigen Isoform p2psa and Its Derivates, %p2psa and Prostate Health Index in the Detection of Prostate Cancer and in Predicting Aggressive Disease: a Prospective Study
Brief Title: Predictive Value of Prostate-specific Antigen Isoform p2psa and Its Derivates in the Diagnosis of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Luigi Mearini, Dr, University Of Perugia
Other Study IDs: propsa12
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer, PSA, markers, diagnosis, prognosis, pro-PSA
MeSH Terms: conditions — Prostatic Neoplasms; Salivary Gland Adenoma, Pleomorphic; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In Europe, prostate cancer (PCa) is the most common solid neoplasm, with an incidence rate of 214 cases per 1000 men, outnumbering lung and colorectal cancer. Early detection tests have been developed in order to identify PCa while it is still confined to the prostate gland.

The two most commonly used tests are digital rectal examination and serum prostate-specific antigen (PSA) level: however, most of cases is detected in the so called T1c stage, i.e. for PSA increasing only. As marker, PSA is organ-specific but not cancer-specific, and its levels may change as result of physical activity, sexual activity, in the presence of benign prostatic hyperplasia (BPH), acute and chronic prostatitis, as well as in the presence of PCa.

A total serum PSA of 4.0 ng/ml has traditionally been used as threshold for considering prostate biopsy and large programs for the early detection of prostate cancer have shown that almost 70% of cancer cases can be detected using a PSA cutoff of 4.0 ng/ml. However, using a PSA threshold of 4.0 ng/ml 20% to 25% of prostate cancer cases are not detected (false-negative) and the false-positive rate is 65%. To improve the usefulness of PSA for identifying patients who require biopsy, the PSA threshold has been lowered at 2 ng/ml; moreover, the levels of free and bound PSA have been assessed, together with PSA density (the rate of PSA over the prostate volume) and PSA velocity (the rate of PSA increase), which seem to have some validity for detecting prostate cancer.

Recent studies have shown that other new biomarkers could be used in the diagnosis of early prostate cancer as they showed a higher sensitivity and specificity. In the last two years, several investigators showed that PSA isoform [-2] proPSA (p2PSA) and its derivatives, namely, percentage of p2PSA to free PSA (%p2PSA) and the Prostate Health Index [PHI; (p2PSA / free PSA) × √tPSA)] improve the accuracy of total PSA (tPSA) and percentage of free PSA (%fPSA) in predicting the presence of PCa at prostate biopsy and they are also related to PCa aggressiveness at biopsy.

The aim of this study is to confirm the diagnostic and prognostic predictive value of prostate-specific antigen isoform p2psa and its derivates, %p2psa and prostate health index in the detection of prostate cancer in patients with a PSA 2-10 ng/ml and/or suspicious DRE.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-75
* Total serum PSA of 2.0-10 ng/ml at entry and/or suspicious digital rectal examination
* Patients suitable for prostate biopsy

Exclusion Criteria:

* History of PCa
* Previous prostate biopsy or prostatic surgery
* History of acute urinary retention within 3 months prior
* Use of any investigational or marketed 5ARI, anabolic steroids or any drug with anti-androgenic properties within 12 months prior to screening.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urological outpatient clinics of one tertiary university high volume department of urology
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
diagnosis of prostate cancer | 6 months
  Analyzing the predictive value of %p2PSA and PHI in comparison with standard test (tPSA, fPSA, %fPSA, PSA density, DRE) in the diagnosis of prostate cancer.

SECONDARY OUTCOMES:
prognosis of prostate cancer | 6 months
  Analyzing the predictive value of %p2PSA and PHI in comparison with standard test (tPSA, fPSA, %fPSA, PSA density, DRE) in the evaluation of aggressiveness of prostate cancer, based on Gleason score groups at biopsy (low risk 4-6, Intermediate risk =7, high risk >=8).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Perugia - Urology Dept, Perugia, Italy